CLINICAL TRIAL: NCT04752735
Title: Endovascular treatmenT for Acute Ischemic Stroke in China: a Retrospective, National, Multi-center, Registry Study
Brief Title: Endovascular treatmenT for Acute Ischemic Stroke in China
Acronym: DETECT-China
Status: Completed | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Head of Neurology, General Hospital of Shenyang Military Region
Other Study IDs: y (2021)013
Record Dates: First submitted 2021-02-10; First posted 2021-02-12 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Stroke; Endovascular Treatment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: endovascular treatment — all enrolled patients must receive endovascular treatment.

SUMMARY:
This is a retrospective real world registry study, aiming to explore the effectiveness and safety of endovascular treatment of acute ischemic stroke in a Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18;
* Ischemic stroke confirmed by head CT or MRI;
* Patients receiving endovascular treatment;
* First ever stroke or mRS≤2 after previous disease;
* Complete and clear pre- and post-operative DSA images are available

Exclusion Criteria:

* Imaging data not qualified for evaluation;
* Absence of important clinical data;
* The first 50 patients receiving endovascular treatment in a single centerr.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients must receive endovascular treatment regardless of the time from onset to treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Score (mRS) 0 to 2 | Day 90
  the minimum and maximum values of mRS are 0 and 6, respectively; higher mRS mean a worse outcome

SECONDARY OUTCOMES:
Changes in National Institute of Health stroke scale (NIHSS) | Day 2, 7, 14
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome
Proportion of patients with modified Rankin Score 0 to 2 | Day180, 360
  Proportion of patients with modified Rankin Score 0 to 2
Distribution of modified Rankin Score | Day 90, 180, 360
  Distribution of modified Rankin Score after treatment
Proportion of symptomatic intracranial hemorrhage (sICH) | 48 hours
  sICH was defined as 4 or more increase in NIHSS caused by hemorrhage
Proportion of intraparenchymal hemorrhage (PH1 and PH2) | 48 hours
  Proportion of intraparenchymal hemorrhage (PH1 and PH2) after treatment
Proportion of death | Day 7
  death due to any cause
Changes in cerebral edema | 48 hours, 7 days
  edema is determined by middle shift.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China

REFERENCES:
- [Derived] Xing GP, Li W, Cui C, Zhao ZA, Nguyen TN, Chen HS. Thrombolysis to Recanalization Time Affects the Benefit of Bridging Thrombolysis in Large Vessel Occlusion Patients With Successful Recanalization. CNS Neurosci Ther. 2025 Sep;31(9):e70579. doi: 10.1111/cns.70579. PMID 40947819